CLINICAL TRIAL: NCT07019285
Title: Comparative Effects of High- vs. Moderate Intensity Interval Walking Training on Plasma Volume Variations, Hematological and Muscle-Damage Markers in Overweight/Obese Postmenopausal Women
Brief Title: Interval Training and Plasma Volume Variation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wissal Abassi (Other)
Responsible Party: Sponsor-Investigator, Wissal Abassi, Principal Investigator, High Institute of Sports and Physical Education of Kef
Organization: High Institute of Sports and Physical Education of Kef (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Hematological markers
Record Dates: First submitted 2025-05-26; First posted 2025-06-13 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: Hematologic Tests
Keywords: Hematocrit; Plasma volume variation; Interval walking training; Lactate dehydrogenase; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-intensity intermittent walking training group (Experimental): performed five 6-minute walking bouts at 90-110% of the 6-minute walking test distance (6MWTD) with 6-min of active recovery between repetitions
  Interventions: Behavioral: High intensity interval walking training
- Moderate-intensity intermittent walking training group (Experimental): repeated five 6-minute walking intervals at 60-80% of 6MWTD interspersed with 6 minutes of active recovery between repetition
  Interventions: Behavioral: Moderate-intensity interval walking training
- Control group (No Intervention): No training intervention was intended for the control group.

INTERVENTIONS:
Behavioral: High intensity interval walking training — High intensity intermittent walking training for a period of 8 weeks. The intensity of the training is 90 to 110% of 6MWTdistance. The frequency of the training is three times a week
  Arms: High-intensity intermittent walking training group
Behavioral: Moderate-intensity interval walking training — Moderate intensity intermittent walking training for a period of 8 weeks. The intensity of the training is 60 to 80% of 6MWTdistance. The frequency of the training is three times a week
  Arms: Moderate-intensity intermittent walking training group

SUMMARY:
The goal of this clinical trial is to to compare the effects of high (HIIWT) versus moderate-intensity interval walking training (MIIWT) on body composition, plasma volume variations (PVV), hematological parameters, muscle damage and aerobic capacity in overweight/obese postmenopausal women. The main question it aims to answer is:Does HIIWT and MIIWT improve kidney function markers in this population? Researchers will compare HIIWT to MIIWT and to non-training intervention(designed to control group) to see if the training program at different intensities work to improve kidney function markers.

Participants in HIIWT group will: perform a 8-week HIIWT program, three sessions per week (5 repetitions of 6-min-walking-test (6MWT) at 90-110% of 6MWTdistance measured at baseline, interspersed by 6-min of active recovery between repetitions). Participants in MIIWT group will: perform a 8-week MIIWT program, three sessions per week (5 repetitions of 6-min-walking-test (6MWT) at 60-80% of 6MWTdistance measured at baseline, interspersed by 6-min of active recovery between repetitions). Participants in control group will : not perform any physical training and maintain their usual daily activities.

DETAILED DESCRIPTION:
In obese postmenopausal women, hematological disturbances, reduced plasma volume, and elevated muscle damage biomarkers are associated with impaired oxygen delivery, reduced aerobic capacity, and increased risks of cardiovascular disease, sarcopenia, and functional decline. While responses to exercise are well documented in young healthy individuals, evidence in this high-risk population remains scarce. The purpose is to compare the effects of high (HIIWT) versus moderate-intensity interval walking training (MIIWT) on body composition, plasma volume variations (PVV), hematological parameters, muscle damage and aerobic capacity in overweight/obese postmenopausal women.Thirty-two overweight/obese postmenopausal women were randomly assigned to HIIWT (n = 11), MIIWT (n = 11), or control (CON, n = 10) groups. HIIWT and MIIWT groups performed intermittent walking at 90-110% and 60-80% of the 6-min-walking-test distance, respectively, 3 times/week for 8 weeks (60 min/session). Body composition, hematological and muscle damage markers, and 6 min walk test (6MWT) were assessed pre- and post-intervention. PVV was calculated after eight weeks under third conditions (HIIWT, MIIWT and CON).

ELIGIBILITY:
Inclusion Criteria:

* Age range of 45-59 years.
* Postmenopausal women (cessation of menses for at least 12 consecutive months).
* Body mass index (BMI) ≥ 25 kg/m2.
* Body weight remained constant (±2 kg) during the past 3 months.
* Stable eating habits and physical activity for at least 3 months.
* Sedentary lifestyle (exercise less than 1h/week).

Exclusion Criteria:

* Medical contraindications to physical activity, diagnosed metabolic, hormonal, orthopedic, or cardiovascular conditions.
* Current use of hormone replacement therapy or any prescribed medication.

Ages: 45 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-03-16 (Actual); Study Completion 2025-03-16 (Actual)

PRIMARY OUTCOMES:
Erythrocytes | At baseline and at week 9 (after the eight weeks of the training intervention).
  Blood levels of erythrocytes were collected from a blood sample (5 ml) and analyzed using a multichannel automated hematology analyzer (XN450; Sysmex, Norderstedt, Germany).
Hemoglobin | At baseline and at week 9 (after the eight weeks of the training intervention).
  Blood levels of hemoglobin were collected from a blood sample (5 ml) and analyzed using a multichannel automated hematology analyzer (XN450; Sysmex, Norderstedt, Germany).
Hematocrit | At baseline and at week 9 (after the eight weeks of the training intervention).
  Blood levels of hematocrit were collected from a blood sample (5 ml) and analyzed using a multichannel automated hematology analyzer (XN450; Sysmex, Norderstedt, Germany).
Mean corpuscular volume | At baseline and at week 9 (after the eight weeks of the training intervention).
  Blood levels of mean corpuscular volume were collected from a blood sample (5 ml) and analyzed using a multichannel automated hematology analyzer (XN450; Sysmex, Norderstedt, Germany).
Mean corpuscular hemoglobin content | At baseline and at week 9(after the eight weeks of the training intervention)
  Description: Blood levels of mean corpuscular hemoglobin content were collected from a blood sample (5 ml) and analyzed using a multichannel automated hematology analyzer (XN450; Sysmex, Norderstedt, Germany).
  Time Frame: At baseline and at week 9 (after the eight weeks of the training intervention)
Mean hemoglobin concentration | At baseline and at week 9 (after the eight weeks of the training intervention)
  Blood levels of mean hemoglobin concentration were collected from a blood sample (5 ml) and analyzed using a multichannel automated hematology analyzer (XN450; Sysmex, Norderstedt, Germany).
Creatine kinase | At baseline and at week 9 (after the eight weeks of the training intervention).
  Serum concentrations of creatine kinase are measured from a blood sample (5 ml) using a Beckman Coulter AU480 Chemistry Analyzer (France).
Lactate dehydrogenase | At baseline and at week 9 (after the eight weeks of the training intervention).
  Serum concentrations of lactate dehydrogenase are measured from a blood sample (5 ml) using a Beckman Coulter AU480 Chemistry Analyzer (France).
Plasma volume variations | Plasma volume variations (PVV) was calculated after eight weeks under third conditions (High intensity training, Moderate intensity training and No training intervention [control group] ).
  Plasma volume variations (PVV) was calculated based on measured hematocrit (Ht) and hemoglobin (Hb) values according to the method developed by Dill and Fink (1974).
  %PVV=100 ×[(Hb0/Hb1) ×(100 - Ht1) / (100 - Ht0)] - 1, where 0 is the value measured before training program and 1 is the value measured after training program.
Body weight | At baseline and after eight weeks of the training intervention.
  Body weight (kg) was recorded , with barefoot and lightly dressed subjects, using an electronic scale (Tanita BC-533, Tokyo, Japan).
Height | At baseline and at week 9 (after the eight weeks of the training intervention).
  Height (m) was determined using a standard stadiometer (Holtain Ltd., UK).
Body fat | At baseline and at week 9 (after the eight weeks of the training intervention).
  Body fat (%) was recorded using an electronic scale (Tanita BC-533, Tokyo, Japan).
Body mass index | At baseline and at week 9 (after the eight weeks of the training intervention).
  Body mass index (kg/m²) was calculated as weight (kg) divided by height squared (m²).
Waist circumference | At baseline and at week 9 (after the eight weeks of the training intervention).
  Waist circumference (cm) was measured to the nearest 0.1 cm using a non-deformable anthropometric tape, placed horizontally at the midpoint between the inferior margin of the last palpable rib and the superior border of the iliac crest, with the participant standing upright and breathing normally.

CONTACTS AND LOCATIONS:
Overall Officials: Wissal abassi, Dr, Principal Investigator — Research Unit "Sport Sciences, Health and Movement"(UR22JS01) High Institute of Sport and Physical Education of Kef, University of Jendouba, 7100 Kef, Tunisia.; Antonella MUSCELLA, Professor, Principal Investigator — Department of Biological and Environmental Science and Technologies (DiSTeBA), University of Salento, 73100 Lecce, Italy.
Locations (1):
- High Institute of Sports and Physical Education of Kef, El Kef, Boulifa, Tunisia

IPD SHARING:
Plan to Share IPD: No
For confidentiality reasons, all data from this study are available upon request.